CLINICAL TRIAL: NCT03667391
Title: Taiwan Cohort - Chronic ThromboEmbolic Pulmonary Hypertension Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201709016RIPC
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: The Geodemographics of CTEPH in Taiwan
Keywords: Chronic ThromboEmbolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH) is difficult for numerous reasons and is related with a poor prognosis. In Taiwan, the incidence of CTEPH and its clinical features are unknown. This study aims at evaluating the prevalence, clinical characteristics, and management of CTEPH in a Taiwanese cohort.

Primary objective:

- To investigate the geodemographics of CTEPH in Taiwan

Secondary objectives:

* To characterize the demographics and clinical presentation of patients with CTEPH
* To describe the real-world management and treatment outcome of patients with CTEPH
* To identify the risk factors of CTEPH
* To assess the relationship between risk factors/patients' characteristics and clinical outcomes for CTEPH
* To evaluate the prognosis of CTEPH in Taiwan using survival assessment

ELIGIBILITY:
Inclusion Criteria:

1. Right heart catheterization (RHC) results that are in line with both of the following haemodynamic levels:

   Mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg at rest AND Pulmonary arterial wedge pressure (PAWP) ≤ 15 mmHg
2. Confirmation of CTEPH diagnosis by one of the following as recommended by standard guidelines:

   At least 1 (segmental) perfusion defect(s) in ventilation-perfusion (V/Q) / perfusion scan OR Pulmonary artery obstruction seen by multidetector computed tomography (MDCT) angiography or conventional pulmonary cineangiography.
3. Presence of pulmonary hypertension or evidence of pulmonary thromboembolism after at least 3 months of anticoagulation treatment.

Exclusion Criteria:

* not written informed consent
* not meet inclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with contrast CT image and cardiac echo data and confirmed/suspected as CTEPH can be included in the screening (initial registration). Those who have confirmed diagnosis of CTEPH in expert centers (IRB approved for patient enrollment) will be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the geodemographics of CTEPH in Taiwan | recruiting period two years
  variables of interest also include (1) patients characteristics, such as demographics and medical history; (2) clinical features and diagnosis records, such as risk factors, comorbidities, CTEPH diagnosis data, concomitant conditions; (3) management of CTEPH, including surgery and medication; and (4) clinical outcome including clinical assessment results, survival status, and clinical worsening related to CTEPH.

SECONDARY OUTCOMES:
To characterize the demographics and clinical presentation of patients with CTEPH - To describe the real-world management and treatment outcome of patients with CTEPH - To identify the risk factors of CTEPH - To assess the relationship between risk f | recruiting period two years
  detail information descriptive in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Hsao H Hsu, PhD, Principal Investigator — No.7, Chung Shan S. Rd.（Zhongshan S. Rd.）, Zhongzheng Dist., Taipei City 10002, Taiwan (R.O.C.)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang KM, Wang MT, Tao CW, Wu YJ, Hsu CH, Liao WC, Hsu HH, Lin MC, Tsai FT, Fu YJ, Kuo FY, Cheng CC, Hung CC, Wang HC, Yu CJ, Huang WC. The long-term outcome of chronic thromboembolic pulmonary hypertension: Pulmonary endarterectomy and balloon pulmonary angioplasty. J Chin Med Assoc. 2024 Mar 1;87(3):273-279. doi: 10.1097/JCMA.0000000000001059. Epub 2024 Jan 22. PMID 38252515